CLINICAL TRIAL: NCT03741712
Title: A Phase I/II,Open-Label,Does-Escalation and -Expansion, Safety,Pharmacokinetics and Efficacy Study of SHR2554 Alone or in Combination With SHR3680 in the Treatment of Patients With Metastatic Castration Resistant Prostate Cancer
Brief Title: A Study of SHR2554 Alone or in Combination With SHR3680 in the Treatment of mCRPC
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: According to the available data from the trial，the sponsor determined to terminate this study.
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHR2554-SHR3680-I/II-102
Record Dates: First submitted 2018-10-17; First posted 2018-11-15 (Actual); Last update posted 2021-02-05 (Actual); Status verified 2018-07

CONDITIONS: Prostate Cancer; Castration-resistant Prostate Cancer
Keywords: Castration-resistant Prostate Cancer; SHR2554; SHR3680
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SHR2554 (Experimental): Participants will receive SHR2554 orally
  Interventions: Drug: SHR2554
- SHR2554+SHR3680 (Experimental): Participants will receive SHR2554 combined with SHR3680 orally
  Interventions: Drug: SHR3680; Drug: SHR2554

INTERVENTIONS:
Drug: SHR3680 — Tablet. Specifications of 80mg
  Arms: SHR2554+SHR3680
Drug: SHR2554 — Tablet. Specifications of 50mg and 200mg

SUMMARY:
The aim of this trial is to study the tolerance, pharmacokinetics (PK) and efficacy of SHR2554 alone or in combination with SHR3680 in the treatment of patients with metastatic Castration Resistant Prostate Cancer.

DETAILED DESCRIPTION:
This is a multicenter, open, non-randomized and dose-escalating and -expansion Phase I/II trial and it studies the tolerance, PK and efficacy of SHR2554 alone or in combination with SHR3680 in the treatment of patients with metastatic Castration Resistant Prostate Cancer. The Phase I part is a dose-escalating study including Ia (dose-escalation monotherapy) and Ib (dose-escalation combination therapy). Approximately 18-30 patients in Phase Ia will only receive one of five dose levels of orally SHR2554. Approximately 30~48 patients in Phase Ib trial will receive SHR2554 combined with SHR3680, in which 2~3 different dose levels of SHR2554 will be selected based on the result of the Phase Ia. Phase II part is a dose-expansion study. Primary endpoints of the study are dose-limiting tolerance (DLT), maximum-tolerated dose (MTD) and prostate specific antigen (PSA) response rate.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed prostate cancer;
2. Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) of 0 or 1;
3. Radiographic evidence of metastasis;
4. Sustained therapy of luteinizing hormone-releasing hormone analogue（LHRHA）or received bilateral orchiectomy; patients who did not receive bilateral orchiectomy are willing to receive sustained therapy of LHRHA;
5. Evidence of prostate cancer progression under the sustained therapy of LHRHA or bilateral orchiectomy;
6. Adequate hepatic, renal, heart, and hematological functions;
7. Patients have given voluntary written informed consent before performance of any study-related procedure not part of normal medical care,with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care.

Exclusion Criteria:

1. Have received any anti-tumor therapy in the past 4 weeks,including radiotherapy, chemotherapy, operation, targeted therapy, immunotherapy, and endocrinotherapy;
2. Planned to initiate any other anti-tumor therapies during the study;
3. Unable to swallow, chronic diarrhea and intestinal obstruction, or the presence of a variety of other factors that affect drug use and absorption;
4. Clinically significant cardiovascular diseases;
5. History of seizure or certain conditions that may predispose to seizure;
6. Severe concurrent disease and infection that, in the judgment of the investigator, would make the patient inappropriate for enrollment.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2018-11-20 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2020-12-08 (Actual)

PRIMARY OUTCOMES:
DLT | Approximately 12 months
  A DLT is any of the predefined set of unacceptable adverse events observed and at least possibly related to investigational agents
MTD | Approximately 12 months
  The first cycle DLTs will be utilized to determine the MTD and future dose escalations or de-escalations The first cycle DLTs will be utilized to determine the MTD and future dose escalations or de-escalations
PSA response rate | Approximately 12 weeks
  After the continuous therapy from randomisation to the end of the 12 weeks, the ratio of patients whose levels of PSA decreased more than 50%

SECONDARY OUTCOMES:
Time to PSA progression | Approximately 70 months
  Time from randomisation to the first time of PSA progression according to the criteria of the Prostate Cancer Clinical Trials Working Group 3 （PCWG3)
Objective response rate (ORR) | Approximately 70 months
  The percentage of subjects with measureable disease at baseline who achieved a complete or partial response in their soft tissue disease using the Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 criteria
Under the Curve (AUC) | Approximately 12 months
  The single dose and multiple dose PK will be calculated as data permits including Area AUC
Maximum Observed Plasma Concentration (Cmax) | Approximately 12 months
  The single-dose and multiple dose PK will be calculated as data permits including Cmax
Adverse events (AE) | Approximately 70 months
  The type, frequency, severity, timing, seriousness, and relationship to study therapy

CONTACTS AND LOCATIONS:
Overall Officials: Dingwei Ye, M.D., Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China